CLINICAL TRIAL: NCT00447265
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase II, Multi-Center Study for Treatment of Lupus Nephritis by Inhibition of Tumor Necrosis Factor-alpha Using Etanercept
Brief Title: Etanercept for the Treatment of Lupus Nephritis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The perceived risk-benefit ratio for individuals with early active RA
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DAIT ALN01
Record Dates: First submitted 2007-03-12; First posted 2007-03-14 (Estimated); Results first posted 2011-12-19 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-02

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis | interventions — Etanercept

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- Etanercept (Experimental): Participants in this group will self-administer 50 mg etanercept injections once a week for 24 weeks. They will continue receiving their usual treatment with corticosteroids and either mycophenolate mofetil (MMF), mycophenolic acid, or azathioprine (AZA).
  Interventions: Drug: Etanercept; Drug: Lupus Treatment- Standard of Care
- Placebo (Placebo Comparator): Participants in this group will self-administer 50 mg placebo injections once a week for 24 weeks. They will continue receiving their usual treatment with corticosteroids and either mycophenolate mofetil (MMF), mycophenolic acid, or azathioprine (AZA).
  Interventions: Drug: Lupus Treatment- Standard of Care; Drug: Placebo

INTERVENTIONS:
Drug: Etanercept — 1.) Immune suppressant. 2.) Tumor necrosis factor (TNF) inhibitor.
  Other Names: Enbrel
  Arms: Etanercept
Drug: Lupus Treatment- Standard of Care — Individualized standard of care treatment for lupus with corticosteroids and with mycophenolate mofetil (MMF), mycophenolic acid, or azathioprine (AZA)
Drug: Placebo
  Arms: Placebo

SUMMARY:
Systemic lupus erythematosus (SLE) is a chronic, multisystem, autoimmune disease in which the body's immune system attacks its own normal tissues. This abnormal autoimmune response can result in damage to many parts of the body, including the skin, joints, lungs, heart, brain, intestines, and kidneys. Kidney problems occur in 60-75 % of lupus patients. The development of lupus-related kidney disease (called lupus nephritis) is associated with an overall worse prognosis.

SLE is usually treated with drugs that try to block inflammation caused by the immune system. These treatments can create their own problems and they do not cure lupus. The drugs that are often used to treat lupus nephritis include prednisone (steroids), cyclophosphamide (Cytoxan), azathioprine (AZA or Imuran), and mycophenolate mofetil (MMF or Cellcept). The main purpose of this study is to evaluate the safety and tolerability of etanercept compared to placebo in combination with standard of care to treat individuals with active lupus nephritis.

DETAILED DESCRIPTION:
Kidney problems associated with lupus nephritis range from asymptomatic protein in the urine to rapidly progressive glomerulonephritis, leading to end-stage renal disease. The goal of therapies is to control kidney manifestations in order to avoid kidney failure, the occurrence of other medical problems and death.

The treatment of lupus nephritis remains problematic. Despite the use of currently available therapies, patients experience disease relapse. Over time, patients develop significant morbidity from the disease as well as from medications used for treatment.

Etanercept, a TNF inhibitor, is proposed as a potential treatment for lupus nephritis. TNF increases the number of reactive B and T cells. TNF levels can be elevated in lupus. Etanercept is believed to work by blocking inflammation, and it is hoped that it will lessen the signs and symptoms of lupus-related kidney disease.

The purpose of this study is to evaluate the safety and tolerability of etanercept compared to placebo in combination with standard therapy to treat individuals with mild or moderately active lupus nephritis.

This study will last 1 year. Participants will be randomly assigned to receive either etanercept or placebo in addition to their regular medications. Participants will self-administer 50 mg etanercept or placebo injections once a week. They will continue receiving their usual treatment with corticosteroids and either MMF, Mycophenolic Acid, or AZA. Treatment with study medication will occur for 24 weeks.

There will be a screening visit followed by a randomization visit, where subjects will receive and learn how to administer the study drug. Subjects will come to the clinic for 9 study visits. A physical exam and blood and urine collection will occur at most study visits. Participants will also be asked to complete a questionnaire on their health at most study visits. Subjects will be contacted by phone 5 times during the 24-week period to assess for adverse events and worsening disease status.

ELIGIBILITY:
Inclusion Criteria:

* Meets at least 4 of the 11 American College of Rheumatology (ACR) 1982 Revised Criteria for the Classification of SLE
* Active lupus nephritis
* Currently has antibodies to double-stranded DNA (dsDNA)
* Currently receiving treatment consisting of at least 1.5 g/day of MMF OR at least 720 mg/day orally of Mycophenolic Acid OR at least 1.5 mg/kg once per day of AZA for lupus nephritis, for at least 28 days prior to study entry
* Stable medication regimen for at least 4 weeks prior to study entry
* Able and willing to self-administer study drug OR has a designated caregiver at home to administer study drug injections
* Willing to use acceptable forms of contraception for the duration of the study

Exclusion Criteria:

* Moderately severe anemia
* Neutropenia
* Thrombocytopenia
* Blood creatinine levels greater than 3.0 mg/dl
* Positive PPD without ongoing treatment for at least 30 days prior to study entry
* Pulmonary fibrotic changes
* Active infections (e.g., HIV, hepatitis B virus [HBV], hepatitis C virus [HCV]) and/or serologic evidence of prior exposure to hepatitis B
* Received a live vaccine within 3 months prior to study entry
* Doubled serum creatinine levels within the 3 months prior to study entry OR end-stage kidney disease
* Dialysis-dependent end-stage kidney disease or membranous nephritis
* History of cancer. Individuals with a history of cervical carcinoma in situ and resected basal and squamous cell carcinomas of the skin are not excluded.
* Receiving prednisone greater than 20 mg/day or equivalent corticosteroid treatment
* Pulse intravenous methylprednisolone within 30 days prior to study entry
* Receiving immunosuppressive agents other than prednisone, MMF, Mycophenolic Acid, AZA, or hydroxychloroquine
* Oral or intravenous cyclosporine, leflunomide IVIG, or plasmapheresis within 3 months prior to study entry
* Current or previous cyclophosphamide treatment
* Use of other experimental agent within 90 days prior to study entry
* Severe, progressive, or uncontrolled kidney, liver, blood, stomach, lung, heart, or brain disease. Individuals with any of these conditions that are related to active SLE are not excluded.
* Previous use of rituximab within 12 months prior to study entry
* Previous or current exposure to any of the following: etanercept (Enbrel), adalimumab (Humira), infliximab (Remicade), or anakinra (Kineret)
* Meets New York Heart Association classification of congestive heart failure (CHF) Class III or greater
* History of myocardial infarction or ischemia
* Current or history of substance abuse
* Known hypersensitivity to any component of the study drug
* Poorly controlled or advanced diabetes mellitus
* History of multiple sclerosis, transverse myelitis, optic neuritis, or epilepsy
* History of noncompliance with other therapies
* Pregnancy or breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-02; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Dall'Era, MD, Study Chair — Division of Rheumatology, University of California, San Francisco; David Wofsy, MD, Study Chair — Department of Medicine, University of California, San Francisco
Locations (6):
- United States (6):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California at San Francisco, San Francisco, California
  - University of Colorado Health Sciences Center, Aurora, Colorado
  - Feinstein Institute for Medical Research NS-L1J Health System, Manhasset, New York
  - University of Rochester, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina

REFERENCES:
- [Background] Aringer M, Graninger WB, Steiner G, Smolen JS. Safety and efficacy of tumor necrosis factor alpha blockade in systemic lupus erythematosus: an open-label study. Arthritis Rheum. 2004 Oct;50(10):3161-9. doi: 10.1002/art.20576. PMID 15476222
- [Background] De Rycke L, Baeten D, Kruithof E, Van den Bosch F, Veys EM, De Keyser F. The effect of TNFalpha blockade on the antinuclear antibody profile in patients with chronic arthritis: biological and clinical implications. Lupus. 2005;14(12):931-7. doi: 10.1191/0961203305lu2240rr. PMID 16425572
- [Background] Mor A, Bingham CO 3rd, Barisoni L, Lydon E, Belmont HM. Proliferative lupus nephritis and leukocytoclastic vasculitis during treatment with etanercept. J Rheumatol. 2005 Apr;32(4):740-3. PMID 15801034
- [Background] Scheinfeld N. A comprehensive review and evaluation of the side effects of the tumor necrosis factor alpha blockers etanercept, infliximab and adalimumab. J Dermatolog Treat. 2004 Sep;15(5):280-94. doi: 10.1080/09546630410017275. PMID 15370396

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant recruitment occurred at 6 sites. All sites were affiliated with a university and utilized a lupus clinic and outside referrals for recruitment. The first site (UCSF) was activated on 1 Feb 2008. The remaining 5 sites (Feinstein, Rochester, Colorado, Duke, and UAB) were activated over the next year.
Pre-assignment Details: The participant signed an informed consent before study screening procedures commenced to assess eligibility criteria (lupus diagnosis with active nephritis, positive ANA, presence of dsDNA antibodies, and stable medication regimens of either mycophenolate mofetil (MMF, CellCept®, Myfortic®) or azathioprine at the screening visit.
Groups:
- Etanercept: Participants (or their caretaker) would administer 50 mg etanercept subcutaneous injections once weekly for 24 weeks. They would continue receiving their usual treatment with corticosteroids and either mycophenolate mofetil or azathioprine.
- Placebo: Participants (or their caretaker) would administer 50 mg placebo subcutaneous injections once weekly for 24 weeks. They would continue receiving their usual treatment with corticosteroids and either mycophenolate mofetil or azathioprine.
Period: Overall Study
Arm/Group | Etanercept | Placebo
Started | 1 | 0
Completed | 0 (The participant completed treatment and discontinued follow-up at week 39 after randomization) | 0
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Etanercept: Participant self-administered 50 mg etanercept subcutaneous injections once weekly for 24 weeks. She continued receiving her usual treatment with corticosteroids and mycophenolate mofetil.
Arm/Group | Etanercept
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Region of Enrollment [Number; unit: Participants]
  United States | 1
Day 0 GFR (mL/min per 1.73m^2) [Mean (Full Range); unit: mL/min/1.73m^2] — Glomerular filtration rate (GFR) is calculated based on the "Modification of Diet in Renal Disease" equation (Levy, AS, Coresh J, Galk E et al, National Kidney Foundation practice guidelines for chronic kidney disease: evaluation, classification, and stratification. Ann Intern Med, 139(2): 137-47, 2003)
  mL/min/1.73m^2 | 96.9 [96.9 to 96.9]
Day 0 random urine protein [Mean (Full Range); unit: mg/dL] | 141 [141 to 141]
SLEDAI total score [Mean (Full Range); unit: Score] — The Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) is a concise measure of lupus disease activity with excellent test-retest reliability and high responsiveness to clinically important changes in the disease. The total score is derived from ratings on 24 conditions plus the Physician's Global Assessment; 0 indicates inactive disease and the maximum theoretical score is 105 with higher scores representing increased disease activity.
  Score | 22 [22 to 22]

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events (AEs)Grade 3 or Higher Experienced by Participant During Treatment Phase of Study
Description: Number of adverse events (AEs) or serious adverse events (SAEs) Grade 3 or higher experienced by participant over the duration of the treatment period. [1]
  [1] This study graded the severity of AEs experienced by the study participant according to the criteria set forth in the National Cancer Institute's Common Terminology Criteria for Adverse Events Version 3.0.
Time Frame: 24 Weeks
Measure: Number; unit: Events
Groups:
- Etanercept: Etanercept plus standard of care
Arm/Group | Etanercept
Number analyzed (Participants) | 1
Events | 0

2. Secondary Outcome: Number of Participant Adverse Events (AEs) From Baseline to Early Study Withdrawal Visit
Description: Number of participant AEs during the trial. This study graded the severity of AEs experienced by the study participant according to the criteria set forth in the National Cancer Institute's Common Terminology Criteria for Adverse Events Version 3.0.
Time Frame: 39 Weeks
Measure: Number; unit: Events
Arm/Group | Etanercept
Number analyzed (Participants) | 1
Events | 3

3. Secondary Outcome: Percent of Participants Who Achieved a Renal Response at Week 24
Description: Percent of study participants who achieved a renal response at 24 weeks.[1]
  [1]A renal response is defined as: 1) 50% reduction in proteinuria compared to baseline as measured by urinary protein: creatinine ratio; and 2) stable or improving renal function as defined by the Glomerular filtration rate (GFR) calculated based on the "Modification of Diet in Renal Disease" equation (Levy, AS, Coresh J, Galk E et al, National Kidney Foundation practice guidelines for chronic kidney disease: evaluation, classification, and stratification. Ann Intern Med, 139(2): 137-47, 2003)
Time Frame: Week 24
Measure: Number; unit: Percent of Participants
Arm/Group | Etanercept
Number analyzed (Participants) | 1
Percent of Participants | 100

4. Secondary Outcome: Time to Participant's Renal Response
Description: Time to when participant achieved a renal response[1]
  [1]A renal response is defined as: 1) 50% reduction in proteinuria compared to baseline as measured by urinary protein: creatinine ratio; and 2) stable or improving renal function as defined by the Glomerular filtration rate (GFR) calculated based on the "Modification of Diet in Renal Disease" equation (Levy, AS, Coresh J, Galk E et al, National Kidney Foundation practice guidelines for chronic kidney disease: evaluation, classification, and stratification. Ann Intern Med, 139(2): 137-47, 2003)
Time Frame: First 24 Weeks of Study Period
Measure: Number; unit: Weeks
Arm/Group | Etanercept
Number analyzed (Participants) | 1
Weeks | 24

5. Secondary Outcome: Participant Systematic Lupus Erythematosus Disease Activity Index (SLEDAI) Score at Baseline and at Early Study Withdrawal Visit
Description: Reported here is the baseline and week 39 Systematic Lupus Erythematosus Disease Activity Index (SLEDAI) scores. The SLEDAI is a concise measure of lupus disease activity with excellent test-retest reliability and high responsiveness to clinically important changes in the disease. The total score is derived from ratings on 24 conditions plus the Physician's Global Assessment; 0 indicates inactive disease and the maximum theoretical score is 105, with higher scores representing increased disease activity.
Time Frame: Baseline, Week 39 (Early Study Withdrawal Visit)
Measure: Number; unit: Points on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 1
Points on a scale
  Baseline SLEDAI Score | 22
  Week 39 SLEDAI score | 8

6. Secondary Outcome: Number of Participants With a C to B Score Change From Baseline to Week 24 in the British Isles Lupus Assessment Group (BILAG) Mucocutaneous Score
Description: Reported here is the number of participants with a change in their BILAG Mucocutaneous Score from C (at baseline) to B (at week 24). A single alphabetic score (A through E) is used to denote disease severity. The BILAG score is a converted numerical score (A=9, B=3, C=1, D=0, E=0). A maximum mucocutaneous score of 9 signifies higher disease activity and a score of 0 is indicative of inactive systematic lupus erythematosus (SLE) in the specified organ system.
Time Frame: Baseline, Week 24
Measure: Number; unit: Participants
Arm/Group | Etanercept
Number analyzed (Participants) | 1
Participants | 1

7. Secondary Outcome: Number of Participants With a B to D Change From Baseline to Week 24 in the British Isles Lupus Assessment Group (BILAG) Musculoskeletal Score
Description: Reported here is the number of participants with a change in their BILAG Musculoskeletal Score from B (at baseline) to D (at week 24). A single alphabetic score (A through E) is used to denote disease severity. The BILAG score is a converted numerical score (A=9, B=3, C=1, D=0, E=0).A maximum musculoskeletal score of 9 signifies higher disease activity and a score of 0 is indicative of inactive systematic lupus erythematosus (SLE) in the specified organ system.
Time Frame: Baseline, Week 24
Measure: Number; unit: Participants
Arm/Group | Etanercept
Number analyzed (Participants) | 1
Participants | 1

8. Secondary Outcome: Number of Participants With an A to B Score Change From Baseline to Week 24 in the British Isles Lupus Assessment Group (BILAG) Renal Score
Description: Reported here is the number of participants with a change in their BILAG Renal Score from A (at baseline) to B (at week 24). A single alphabetic score (A through E) is used to denote disease severity. The BILAG score is a converted numerical score (A=9, B=3, C=1, D=0, E=0).A maximum renal score of 9 signifies higher disease activity and a score of 0 is indicative of inactive systematic lupus erythematosus (SLE) in the specified organ system
Time Frame: Baseline, Week 24
Measure: Number; unit: Participants
Arm/Group | Etanercept
Number analyzed (Participants) | 1
Participants | 1

9. Secondary Outcome: Participant Medical Outcome Study Short-Form 36 (SF-36) Physical Component Score at Baseline and Week 24
Description: Reported here is the participant baseline and week 24 SF-36 Physical Component scores. The SF-36 measures 8 domains: physical functioning, role limitations due to physical health, body pain, social functioning, mental health, role limitations due to emotional problems, vitality, and general health perceptions[1]. The Physical Component scores of the SF-36 range from 0 to 100; 0 equals worst health state. Higher numbers reported here indicate more improvement in condition from baseline.
  [1]Ref: Ware JE, Sherbourne CD. The MOS36-item short-form health survey Med Care. 1992; 30:473-483.
Time Frame: Baseline, Week 24
Measure: Number; unit: Score on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 1
Score on a scale
  Baseline SF-36 Physical Component Score | 44.4
  Week 24 SF-36 Physical Component Score | 42.3

10. Secondary Outcome: Participant Medical Outcome Study Short Form 36 (SF-36) Mental Component Score at Baseline and Week 24
Description: Reported here are the participant SF-36 Mental Component scores at baseline and week 24. The SF-36 measures 8 domains: physical functioning, role limitations due to physical health, bodily pain, social functioning, mental health, role limitations due to emotional problems, vitality, and general health perceptions.[1] The Mental Component score of the SF-36 ranges from 0 to 100; 0 equals worst health state. Higher numbers reported here indicate more improvement in condition from baseline.
  [1]Ref: Ware JE, Sherbourne CD. The MOS36-item short-form health survey. Med Care. 1992; 30:473-483
Time Frame: Baseline, Week 24
Measure: Number; unit: Score on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 1
Score on a scale
  Baseline SF-36 Mental Component Score | 31.4
  Week 24 SF-36 Mental Component Score | 52.3

ADVERSE EVENTS:
Time Frame: Baseline to 39 weeks
Description: This study graded the severity of adverse events experienced by the study participant according to criteria set forth in the National Cancer Institute's Common Terminology Criteria for Adverse Events Version 3.0
Groups:
- Etanercept: Participant received self-administered 50 mg etanercept subcutaneous injections once weekly for 24 weeks while continuing to receive her usual lupus treatment of corticosteroids and mycophenolate mofetil.
Arm/Group | Etanercept
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etanercept (N=1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Muscle Strain (Injury, poisoning and procedural complications) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)

LIMITATIONS AND CAVEATS:
The study terminated early with 1 subject enrolled. Based on safety info from other trials, the protocol chairs decided possible risks to patients outweighed the potential benefits. Analysis of groups is not possible. Study objectives cannot be met.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No